CLINICAL TRIAL: NCT02118506
Title: Immediate Effects of Mental Practice in Gait of Individuals With Parkinson Disease: Randomized Clinical Trial
Brief Title: Effects of Mental Practice in Gait of Individuals With Parkinson Disease: Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Ana Raquel Rodrigues Lindquist, PhD Ana Raquel Rodrigues Lindquist, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CEP/UFRN 275.155
Record Dates: First submitted 2014-01-20; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson Disease
Keywords: Primary Parkinsonism.; Rehabilitation.; Biomechanics.; Neurological gait disorders.
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical practice (Active Comparator): Familiarization with gait cycle: Cards with pictures of an elderly person performing movements related to the adjustment of posture, gait initiation and gait phases were shown to the subjects. They should have organized them sequentially, showing that they learned gait phases.
  Physical practice: is the execution of the motor action.
  Interventions: Other: Physical practice
- Mental and physical practice (Experimental): Familiarization with gait cycle: Cards with pictures of an elderly person performing movements related to the adjustment of posture, gait initiation and gait phases were shown to the subjects. They should have organized them sequentially, showing that they learned gait phases.
  Mental practice: is defined as motor imagery training with the aim of improving the engine performance. Is the imagination of a motor action without its physical implementation.
  Physical practice: is the execution of the motor action.
  Interventions: Other: Mental and physical practice

INTERVENTIONS:
Other: Physical practice — The control group underwent familiarization of gait phases using cards with gait phases and physical gait training.
  Familiarization with gait cycle: Cards with pictures of an elderly person performing movements related to the adjustment of posture, gait initiation and gait phases were shown to the subjects. They should have organized them sequentially, showing that they learned gait phases. Then, they were submitted to a physical gait training. They underwent a single training session during 1 hour and 30 minutes and were reassessed 10 minutes and 1 day after the end of the session, in respect of the kinematic gait and mobility.
  Arms: Physical practice
Other: Mental and physical practice — The experimental group underwent familiarization of gait phases using cards with gait phases, mental practice of gait and physical gait training.
  Familiarization with gait cycle: Cards with pictures of an elderly person performing movements related to the adjustment of posture, gait initiation and gait phases were shown to the subjects. They should have organized them sequentially, showing that they learned gait phases.
  Then, they were submitted to a mental training of gait. They imagined the gait steps per 400 repetitions. While imagining, they verbalized the gait phases.
  Finally, they were submitted to a physical gait training. They executed 400 steps.
  They underwent a single training session during 1 hour and 30 minutes and were reassessed 10 minutes and 1 day after the end of the session, in respect of the kinematic gait and mobility.
  Arms: Mental and physical practice

SUMMARY:
The purpose of this study is to compare the effects of mental practice, associated with physical practice, on gait (cinematic parameters and mobility) in individuals with idiopathic Parkinson's disease. It is believed that familiarity with the normal gait pattern, associated with mental practice and physical practice can trigger significant changes in spatiotemporal and angular parameters that are not observed in the group not submitted to mental practice.

ELIGIBILITY:
Inclusion Criteria:

* the subjects should be in use of antiparkinsonian medication,
* be between stages 2 and 3 of the Hoehn and Yahr modified scale);
* walk without any brace or aid device, independently (scores between 3 and 5 of the Functional Ambulatory Category - FAC) for at least 10 meters
* were not undergoing stereotactic surgery.

Exclusion Criteria:

* We excluded those who were unable or declined to complete the training protocol.

Ages: 44 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Step length at 10 minutes and 1 day | Three observetions were done. At baseline, 10 minutes and 1 day after intervention.

SECONDARY OUTCOMES:
Change from Baseline in Double Limb Support Time at 10 minutes and 1 day | Three observetions were done. At baseline, 10 minutes and 1 day after intervention.
  Double Limb Support Time is the period when both feet are on the ground at the same time. The first period of double limb support begins at initial contact, and lasts, in healthy people, 10 to 12 percent of the cycle. The second period of double limb support occurs in the final 10 to 12 percent of stance phase. As the stance limb prepares to leave the ground, the opposite limb contacts the ground and accepts the body's weight. The two periods of double limb support account for 20 to 24 percent of the gait cycle's total duration. In people with Parkinson disease, this period lasts longer.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenna M. de Melo Santiago, Master, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil